CLINICAL TRIAL: NCT05881499
Title: The Effects of 2023 Earthquakes on Fear of Movement and Fear of Falling in Turkish Survivors: an Observational Cross-sectional Study
Brief Title: The Effects of Earthquake on Fear of Movement and Fear of Falling
Status: Completed | Type: Observational
Sponsor: Nagihan Acet (Other)
Responsible Party: Sponsor-Investigator, Nagihan Acet, Asst. Prof., Atılım University
Organization: Atılım University (Other)
Other Study IDs: Atılım University
Record Dates: First submitted 2023-05-03; First posted 2023-05-31 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2023-11

CONDITIONS: Fear of Movement; Fear of Falling
Keywords: Earthquake; Kinesiophobia
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In February-March 2023, a series of major earthquakes occurred in 11 provinces of Turkey (Adana, Adıyaman, Diyarbakır, Gaziantep, Hatay, Kahramanmaraş, Kilis, Malatya, Osmaniye, Şanlıurfa and Elazığ). The current study is planned as a observational cross-sectional study with the participation of the survivors who experienced the 2023 earthquakes and aftershocks in Turkey without any physical injury during or after the earthquake. It is planned for the participants to fill out the questionnaires by considering the time periods before and after the earthquake. While the primary outcome is fear of movement and fear of falling, the secondary outcome is level of physical activity and intensity of pain. Psychological resilience level was considered as a predictive factor.

The aim of the current study is to determine the effect of earthquake experience on the fear of movement and falling in earthquake victims and to investigate the factors related with them. Fear of movement, fear of falling, level of physical activity, intensity of pain and psychological resilience are evaluated with the Causes of Fear of Movement Scale, Modified Falls Efficacy Scale, Short Form of International Physical Activity Questionnaire, Numerical Pain Scale and Connor-Davidson Psychological Resilience Scale respectively.

DETAILED DESCRIPTION:
INTRODUCTION: Major earthquakes increase the risk of mental and emotional diseases such as anxiety disorders, sleep disorders and post-traumatic stress disorder as well as physical and biological complaints such as dizziness, vertigo and balance disorder.

An elaborate study conducted by Nomura et al., propounded the concept of Post-Earthquake Dizziness Syndrome (PEDS) for dizziness like features in earthquake victims. Their study also indicated that a previous history of vertigo was not related to the prevalence of PEDS. However, they noted that people prone to motion sickness were found to have a significantly higher prevalence of post-earthquake dizziness episodes.

In a previous review study conducted in 2021, the results showed that the prevalence of balance disorders increased significantly after the major earthquakes when compared to before the earthquakes. Exposure to major earthquakes and aftershocks has been shown to cause post-earthquake balance disorders by causing sensory conflicts mediated by vestibular dysfunction and/or psychological factors. In addition, that study stated that this increase in the prevalence of balance disorders may also be caused by psychological factors, which is consistent with previous studies in the literature.

The mechanisms of equilibrium dysfunction are likely to be explained by the sensory conflict theory/postural instability theory. The basic pathology of equilibrium dysfunction is attributed to disruption of interplay between vestibular, neurological, visual and proprioceptive functions of the human body. Psychological stress and maladaptive visual/somatosensory inputs caused by the earthquake may cause changes in the sense of movement, which is an important component of proprioception sense. Moreover, disruptions in the vestibular system may trigger the fear of falling, leading to decreases in physical activity capacity.

Although some previous studies have reported the presence of diziness or equilibrium disorders, in survivors after the earthquake, no study has investigated the fear of movement and fear of falling in these individuals.

Considering Turkey's geographical location in a high-risk seismic zone, determining the prevalence of fear of movement and falling in earthquake-exposed individuals would greatly contribute to the development of a better empirical approach to post-earthquake disaster management.

The primary aim of the present study is to determine the prevalence of fear of movement and falling in post-earthquake victims without physical injury, while the secondary aim is to reveal the relationship between these two parameters, as well as physical activity level, and pain intensity. Psychological resilliance is considered as a predictıve factor.

According to the the results of current study, it will be determined whether earthquake survivorship should be taken into account in preventing physical inactivity and related complications. In cases where this necessity is determined, rehabilitation programs should be revised depending on the earthquake victim's status.

MATERYAL-METHOD Design of the Study The present study is planned as a observational cross-sectional study and it will include victims of the 2023 earthquake in Türkey. Approval will be obtained from the Atılım University Ethics Committee with 02.05.2023 date and E-59394181-604.01.02-60355 number to be determined.

After providing information about the study, participants who voluntarily agree to participate will be included after obtaining written consent.

For the current study, sample selection will be planned with the simple randomization method. The advantages of this method are that it provides a fair chance for each unit in the population to be selected, eliminates potential biases, and allows for statistical inferences to be made.

The data will be collected through communication with local authorities at the aid points located in the earthquake-affected cities. Surveys will be conducted face-to-face with earthquake victims living in different cities.

In this study, participants will answer the questions by considering two different time periods: first considering the three-week period before the earthquake, and then considering the three-week period after the earthquake. The evaluation will be completed when there are no unanswered questions.

Participants The participants in this study will include individuals who meet the following inclusion criteria: they must be victims of the 2023 earthquake in Turkey and be between the ages of 18 and 60.

Exclusion criteria for participation in the study will be the presence of pre-existing cognitive and/or psychological illness, physical injury status after the earthquake, and illiteracy.

Data collection The primary outcomes of this study are fear of movement and fear of falling, while the secondary outcomes are the level of physical activity and intensity of pain. Psychological resilience level is considered as a predictive variable.

These outcomes will be assessed using the Causes of Fear of Movement Scale, Modified Falls Efficacy Scale, Short Form of International Physical Activity Questionnaire, Numerical Pain Scale, and Connor-Davidson Psychological Resilience Scale, respectively.

Sociodemographic characteristics The sociodemographic characteristics of the participants, such as age, height, weight, body mass index, education status, occupation, income status (income-expenditure relationship), presence of chronic diseases, shelter status, and marital status, will be recorded in a descriptive manner.

Assessment of fear of movement: The fear of movement will be assessed using the Turkish version of the Causes of Fear of Movement Scale. This questionnaire, developed by Janusz Kocjan et al. in 2014, consists of 20 questions and aims to diagnose and identify the causes of motor inactivity.

The questionnaire is divided into two parts, biological and psychological, to determine the reasons for the fear of movement. This structure enables the identification of individual causes of kinesiophobia and the determination of biological and psychological causes separately. The total score obtained from the questionnaire is calculated as the average of the scores obtained from the biological and physiological sub-dimensions. In the updated version from 2018, the total score ranges from 0 to 5. The scale uses a 5-point Likert scoring system (1=I totally disagree, 5=I totally agree). A high score indicates a higher level of fear of movement.

Asseement of fear of falling: The Modified Falls Efficacy Scale with 14 items (10 indoor and 4 outdoor activities) will be used to assess fear of falling. It evaluates participants' confidence during different daily tasks and is a reliable and valid scale for estimating balance and mobility problems. The scale includes items scored between 0 (not confident) and 10 (completely confident) to assess participants' self-efficacy levels regarding falling. The scale score is calculated by dividing the sum of the scores per question by the number of questions. High score means that the sense of safety and competence against falling are high. Cronbach's alpha internal consistency coefficient (ICC) of the scale was found to be 0.93. The Turkish version developed by Çetişli-Korkmaz et al. will be used in this study.

Level of Physical Activity: Turkish version of the Short Form of the International Physical Activity Questionnaire is used in order to determine the level of physical activity and sedentary lifestyles.

The durations of physical activities are multiplied by the Metabolic Equivalent of Task (MET) values per activity, and the results of all items are summed to create a total score for overall physical activity. Physical activity levels are classified into three categories: physically inactive (<600 MET min/week), low physical activity level (600-3000 MET min/week), and sufficient physical activity level (>3000 MET min/week).

Intensity of pain: A 10 cm Numerical Pain Scale will be used to determine the severity of pain, with numbers ranging from "0" (no pain) to "10" (unbearable pain).

Psychological Resilience Status: Psychological Resilience Status will be assessed using the Connor-Davidson Resilience Scale (CD-RISC-25). The Turkish version, developed by Karaırmak, consists of 25 questions and three sub-dimensions, namely perseverance and personal competence, tolerance for negative events and spiritual tendency. The first sub-dimension, 'perseverance and personal competence,' has a maximum score of 60, the second sub-dimension, 'tolerance for negative events,' has a maximum score of 24, and the third sub-dimension, 'spiritual tendency,' has a maximum score of 16. The scale uses a 5-point Likert-type scoring system, ranging from 0-4 points, with "never true" (0 points) to "almost always true" (4 points) as response options. The highest possible score is 100 points, indicating a higher level of psychological resilience as the score increases.

Sample size calculation: Sample size will be calculated after a pilot study.

Statistics:

The data collected from the participants will be analyzed using SPSS statistical software. Descriptive statistics such as mean, standard deviation, and frequency distributions will be used to describe the demographic characteristics and study variables. The normality of the distribution of the study variables will be tested using the Shapiro-Wilk test. If the distribution is normal, the paired sample t-test will be used to compare the pre- and post-earthquake scores of fear of movement, fear of falling, intensity of pain, and physical activity level. In case of non-normal distribution, the Wilcoxon signed-rank test will be used for analysis. Additionally, Pearson correlation coefficient analysis will be used to investigate the relationships between fear of movement, fear of falling, intensity of pain, and physical activity level. A significance level of p<0.05 will be used for all statistical tests.

ELIGIBILITY:
Inclusion Criteria:

-being physically uninjured survivors of the 2023 earthquake in Turkey between the ages of 18 and 60

Exclusion Criteria:

* the presence of pre-existing cognitive and/or psychological illness
* physical injury status after the earthquake
* illiteracy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Uninjured survivors of the 2023 earthquake who voluntarily agree to participate will be included. For the current study, sample selection will be planned with the simple randomization method. The data will be collected through communication with local authorities at the aid points located in the earthquake-affected cities. Surveys will be conducted face-to-face with earthquake victims living in different cities.
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Fear of movement | up to one month
  The fear of movement will be assessed using the Turkish version of the Causes of Fear of Movement Scale. The questionnaire is divided into two parts, biological and psychological, to determine the reasons for the fear of movement. This structure enables the identification of individual causes of kinesiophobia and the determination of biological and psychological causes separately. The scale uses a 5-point Likert scoring system (1=I totally disagree, 5=I totally agree). A high score in the questionnaire indicates that the individual has more fear of movement.
Fear of falling | up to one month
  The Modified Falls Efficacy Scale with 14 items (10 indoor and 4 outdoor activities) will be used to assess fear of falling. It evaluates participants' confidence during different daily tasks and is a reliable and valid scale for estimating balance and mobility problems. The scale includes items scored between 0 (not confident) and 10 (completely confident) to assess participants' self-efficacy levels regarding falling. High score means that the sense of safety and competence against falling are high

SECONDARY OUTCOMES:
Level of physical activity | up to one month
  Turkish version of the Short Form of the International Physical Activity Questionnaire wiil be used in order to determine the level of physical activity and sedentary lifestyles.
  The durations of physical activities are multiplied by the Metabolic Equivalent of Task (MET) values per activity, and the results of all items are summed to create a total score for overall physical activity. Physical activity levels are classified into three categories: physically inactive (<600 MET min/week), low physical activity level (600-3000 MET min/week), and sufficient physical activity level (>3000 MET min/week).
Intensity of pain | up to one month
  A 10 cm Numerical Pain Scale will be used to determine the severity of pain, with numbers ranging from "0" (no pain) to "10" (unbearable pain)
Psychological Resilience Status | up to one month
  Psychological Resilience Status will be assessed using the Connor-Davidson Resilience Scale. It consists of 25 questions and three sub-dimensions, namely perseverance and personal competence, tolerance for negative events and spiritual tendency.
  The first sub-dimension, 'perseverance and personal competence,' has a maximum score of 60, the second sub-dimension, 'tolerance for negative events,' has a maximum score of 24, and the third sub-dimension, 'spiritual tendency,' has a maximum score of 16. The scale uses a 5-point Likert-type scoring system, ranging from 0-4 points, with "never true" (0 points) to "almost always true" (4 points) as response options. The highest possible score is 100 points, indicating a higher level of psychological resilience as the score increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)